CLINICAL TRIAL: NCT06003348
Title: Hydroxycitrate: A Novel Therapy for Calcium Phosphate Urinary Stones
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Naim Maalouf, Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-0339
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Calcium Phosphate Kidney Stones
Keywords: Urolithiasis; Calcium phosphate; Citrate; Acid-base
MeSH Terms: conditions — Urolithiasis | interventions — Super Citrimax; Potassium Citrate

STUDY DESIGN:
Intervention Model Description: In this double-blind, placebo-controlled, randomized, crossover study, each participant will undergo 4 phases of study, with the order randomized by a blocked randomization scheme. The 4 phases will be Placebo, Super CitriMax (OHCit) low dose, Super CitriMax (OHCit) standard dose, or Potassium Citrate. Randomization will be stratified based on sex, concomitant thiazide use, and concomitant alkali use.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Potassium Citrate (Urocit®-K) (Active Comparator): Potassium Citrate KCit 10 mEq 2 tabs, twice daily and Placebo 1 tab, twice daily Total Daily Dose: Citrate 40 mEq/d
  Interventions: Drug: Potassium Citrate
- Super CitriMax; OHCit-standard dose (Experimental): Super CitriMax 7 mEq 3 tabs, twice daily Total Daily Dose: OHCit 42 mEq/d
  Interventions: Dietary Supplement: OHCit- standard dose
- Super CitriMax; OHCit-low dose (Experimental): Super CitriMax 7 mEq 2 tabs, twice daily And Placebo 1 tab, twice daily Total Daily Dose: OHCit 28 mEq/d
  Interventions: Dietary Supplement: OHCit- low dose
- Placebo (Placebo Comparator): Placebo 3 tablets twice daily Total Daily Dose: None
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: OHCit- standard dose — Hydroxycitrate Over-the-counter supplement, not FDA approved or regulated.
  Other Names: Super Citrimax
  Arms: Super CitriMax; OHCit-standard dose
Drug: Potassium Citrate — 10 mEq Extended-release tablets for oral use
  Other Names: Urocit®-K
  Arms: Potassium Citrate (Urocit®-K)
Drug: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: OHCit- low dose — Hydroxycitrate Over-the-counter supplement, not FDA approved or regulated.
  Other Names: Super Citrimax
  Arms: Super CitriMax; OHCit-low dose

SUMMARY:
This study tests whether hydroxycitrate, a molecule closely related to citrate, can reduce calcium phosphate stone recurrence.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled, randomized, crossover study, each participant will undergo 4 phases of study, with the order randomized by a blocked randomization scheme. The 4 phases will be Placebo, Super CitriMax (hydroxycitrate) OHCit low dose, OHCit standard dose, or Potassium Citrate. Randomization will be stratified based on sex, concomitant thiazide use, and concomitant alkali use.

Each phase will be 1 week in duration, during which subjects will take assigned study medications. A minimum 1-week washout period will be imposed between phases. During the first 2 days of each phase, subjects will be instructed to adhere to a prescribed diet. On the last 5 days of each phase, subjects will be kept on a constant metabolic diet. Use of metabolic diet is essential to eliminate confounders that could occur from changes in dietary intake across phases. During the final two study days (days 6-7), two 24-hr urines will be collected for urine biochemistry and crystallization studies. Fasting blood will be obtained at the end of the last urine collection.

Study Medications: Subjects will receive three tablets twice daily during each phase. These will consist of either placebo, Potassium Citrate (KCit), or Super CitriMax (OHCit). Study tablets will be prepared by a compounding pharmacy, with placebo tablets similar in appearance and size to the active medication tablets.

ELIGIBILITY:
Inclusion Criteria:

- Calcium Phosphate stone formers

Exclusion Criteria:

* History of recurrent urinary tract infections
* Chronic diarrhea
* Estimated Glomerular Filtration Rate (eGFR) < 45 ml/min/1.73 m2
* History of primary hyperparathyroidism
* Hypokalemia
* Hyperkalemia
* Pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Formation product (FP) for Calcium Phosphate | After 1 week of treatment
  FP is obtained by adding increasing amounts of Calcium Chloride (CaCl2) to a series of urine aliquots maintained at constant pH for 2 hours, and is identified by the point at which calcium phosphate (CaP) precipitates as detected by an absorbance microplate reader.
  Calculated supersaturation using [Calcium] and [Phosphate] at that point represents FP.

SECONDARY OUTCOMES:
Crystal growth of Calcium Phosphate | After 1 week of treatment
  We will assess crystal growth (CG) of CaP after seeding urine with a small amount of brushite (0.25 mg/ml urine) and incubating at 37°C for 3 hours (representing steady state) under constant stirring. A decrement in [Calcium]×[Phosphate] after seeding signifies crystal growth, while a [Calcium]×[Phosphate] increment represents crystal dissolution.
Calcium Phosphate supersaturation | After 1 week of treatment
  Supersaturation of calcium phosphate will be assessed by Joint Expert Speciation System (JESS).

CONTACTS AND LOCATIONS:
Overall Officials: NAIM M MAALOUF, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States